CLINICAL TRIAL: NCT00371618
Title: Comparison of Outcomes of Interventional Pain Management Procedures Performed With or Without Fluoroscopy: A Retrospective Analysis
Brief Title: IPM Procedures With or Without Fluoroscopy: Outcome Comparison
Status: Withdrawn | Type: Observational
Sponsor: Pain Management Center of Paducah (Other)
Other Study IDs: protocol 13
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain; Neck Pain
Keywords: Fluoroscopy; Interventional Pain Management Procedures
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Fluoroscopy

SUMMARY:
To determine clinically significant improvement in the patients undergoing procedures under fluoroscopy.

To evaluate and compare the adverse event profile in both groups

DETAILED DESCRIPTION:
For the target delivery of injectate, it is believed that fluoroscopy is mandatory. However, there is a view among some professionals that a procedure may be performed without fluoroscopy as effectively as under fluoroscopy. The outcomes among the two groups of patients have not been studied

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone the following procedures:

Cervical facet joint nerve blocks, thoracic facet joint nerve blocks, lumbar facet joint nerve blocks, lumbar interlaminar epidural steroid injections, cervical Interlaminar epidural steroid injections

During 1998 to 2001 and 2004 to 2005

-

Exclusion Criteria: Non-availability of appropriate data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: currently enrolled patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1998-01; Study Completion 2004-05

PRIMARY OUTCOMES:
To demonstrate clinically significant improvement in the patients undergoing procedures under fluoroscopy.
To evaluate and compare the adverse event profile in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States